CLINICAL TRIAL: NCT06958757
Title: This RCT Included 64 Participants (18-30y) With PFP, Ankle Dorsiflexion ROM <10°, and BMI 18.5-28 kg/m². Exclusions: Ankle Fractures, Achilles Rupture, Rheumatoid Arthritis, Gout, Systemic Diseases, or Prior Knee/Ankle Surgeries. Randomized to Two Groups (n=32/Group): Experimental (Standard Exercise + Ankle Dorsiflexion Training) vs Control (Standard Exercise Only) at Matched Intensity/Frequency for 8 Weeks. Outcomes: VAS Pain, Kujala Scale, Ankle Dorsiflexion ROM. Certified Physiotherapists Supervise Sessions. Data Analyzed With SPSS 26.0. The Protocol Complies With the Helsinki Declaration.
Brief Title: A Study on the Effectiveness of Ankle Dorsiflexion Range of Motion Training in Patients With Patellofemoral Joint Pain.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tianjin University of Sport (Other)
Responsible Party: Principal Investigator, Wu Yuan, Principal Investigator, Tianjin University of Sport
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TJUS2025-054
Record Dates: First submitted 2025-04-19; First posted 2025-05-06 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-04

CONDITIONS: Patellofemoral Pain, PFP
MeSH Terms: conditions — Patellofemoral Pain Syndrome

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): standard exercise + ankle dorsiflexion training
  Interventions: Other: Standard Exercise Therapy + Ankle Dorsiflexion Training
- control group (Active Comparator): standard exercise only
  Interventions: Other: Standard Exercise Therapy Only

INTERVENTIONS:
Other: Standard Exercise Therapy + Ankle Dorsiflexion Training — The experimental group receives:
  Standard Exercise Therapy (30 min/session, 3x/week for 8 weeks): Quadriceps eccentric exercises (e.g., slow step-downs), Hip abductor strengthening (e.g., side-lying leg lifts), and Neuromuscular control drills (e.g., single-leg balance on unstable surfaces).
  Ankle Dorsiflexion Training (15 min/session, 3x/week for 8 weeks): Mobilization techniques (posterior glides of the talus), Resistance band exercises (dorsiflexion against elastic bands), Progressive Achilles tendon stretching (weight-bearing calf stretches).
  Exercise progression (resistance/intensity) is adjusted biweekly based on functional assessments.
  Arms: experimental group
Other: Standard Exercise Therapy Only — Standard Exercise Therapy (30 min/session, 3x/week for 8 weeks): Quadriceps eccentric exercises (e.g., slow step-downs), Hip abductor strengthening (e.g., side-lying leg lifts), and Neuromuscular control drills (e.g., single-leg balance on unstable surfaces).
  Exercise progression (resistance/intensity) is adjusted biweekly based on functional assessments.
  Arms: control group

SUMMARY:
Patellofemoral Pain (PFP) is a common knee condition causing pain around the kneecap during activities like running or squatting. Limited ankle flexibility ("dorsiflexion" - how far participants can lift their toes toward the shin) may worsen PFP by altering leg movements. This study investigates whether adding ankle flexibility exercises to standard knee-strengthening programs improves outcomes for young adults with PFP. Active adults aged 18-30 with PFP and limited ankle flexibility (measured with a simple tool) are eligible, excluding those with prior knee/ankle surgeries, fractures, or conditions like arthritis. Sixty-four participants will be randomly assigned to either an Exercise + Ankle Training group (standard knee exercises plus targeted ankle training) or an Exercise-Only group for 8 weeks under physiotherapist guidance. Outcomes include improvements in knee pain scores (Kujala Scale), ankle flexibility changes, and muscle coordination measured with non-invasive sensors. If effective, ankle flexibility training could provide a low-cost addition to current treatments, helping patients resume activities with less pain. The study follows international ethical guidelines and has received preliminary ethics approval (No. TJUS-2025-054).

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-30 years
* Diagnosed with patellofemoral pain (PFP) per clinical guidelines (anterior knee pain aggravated by ≥2 activities: running, squatting, stair climbing)
* Ankle dorsiflexion range of motion (ROM) <10° (measured via goniometer in weight-bearing)
* BMI 18.5-28 kg/m²
* Engage in regular physical activity (≥3 sessions/week)

Exclusion Criteria:

* Ankle fractures
* Achilles tendon rupture
* Rheumatoid arthritis
* Gout, or systemic diseases
* Prior knee/ankle surgeries
* Concurrent lower limb injuries (e.g., ligament tears, meniscal pathology)
* Neurological disorders affecting mobility
* Participation in other lower limb rehabilitation programs within 3 months

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 64 (Estimated)
Dates: Start 2025-05-06 (Estimated); Primary Completion 2025-09-10 (Estimated); Study Completion 2025-09-10 (Estimated)

PRIMARY OUTCOMES:
Kujala Anterior Knee Pain Scale | Assess all outcome measures at baseline (pre-intervention) and immediately after the completion of the 8-week intervention program (post-intervention).
Ankle dorsiflexion range of motion | Assess all outcome measures at baseline (pre-intervention) and immediately after the completion of the 8-week intervention program (post-intervention).

SECONDARY OUTCOMES:
sEMG co-contraction ratios | All outcome measures (sEMG co-contraction) ratios are assessed at baseline (pre-intervention) and immediately after completing the 8-week intervention program (post-intervention).

IPD SHARING:
Plan to Share IPD: No